CLINICAL TRIAL: NCT03465631
Title: Distal Upper Extremity Rehabilitation Using SMART Glove System With Transcranial Direct Current Stimulation (tDCS) for Stroke Patients : a Double-blinded, Randomized Controlled Trial
Brief Title: Upper Extremity Rehabilitation Using SMART Glove System With Transcranial Direct Current Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2016-03-026
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Stroke
Keywords: stroke rehabilitation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART Glove system with dual-tDCS (Experimental): VR-based SMART Glove system with dual-tDCS
  Interventions: Device: SMART Glove system with tDCS
- SMART Glove system with sham-tDCS (Sham Comparator): VR-based SMART Glove system with sham-tDCS
  Interventions: Device: SMART Glove system with sham-tDCS

INTERVENTIONS:
Device: SMART Glove system with tDCS — combined bilateral tDCS and VR-based therapy on distal upper extremity training in patients with stroke.
  Arms: SMART Glove system with dual-tDCS
Device: SMART Glove system with sham-tDCS — combined bilateral tDCS and VR-based therapy on distal upper extremity training in patients with stroke.
  Arms: SMART Glove system with sham-tDCS

SUMMARY:
The aim of this study to investigate the effect of combined bilateral tDCS and VR-based therapy on distal upper extremity training in patients with stroke. We hypothesized that experimental group (VR-based training with dual-tDCS) would improve distal upper extremity function rather than control group (VR-based training with dual sham tDCS).

DETAILED DESCRIPTION:
This is a double-blind, randomized controlled study. Patients were randomly assigned to 1 : 1 ratio to experimental group (VR-based training with dual-tDCS; VR-Dual) or the control group (VR-based training with dual sham tDCS; VR-Sham) . For both conditions, VR-Dual and VR-Sham group commenced at the same time (20 minutes). The therapist and patients were blinded as to whether the patients received real or sham tDCS. The study was approved by the Ethics Committee of the National Rehabilitation Center, Korea, and all participants provided written informed consent before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* first-time ischemic or hemorrhagic stroke
* unilateral upper extremity functional deficits after stroke
* presence of a score of at least 3 points on the Medical Research Council (MRC)
* a score ≥ 4 on the Brunnstrom stage
* a score ≥ 25 on the Korean version of the Mini-Mental Status Exam (K-MMSE)

Exclusion Criteria:

* age < 20 years
* wrist and finger spasticity with the Modified Ashworth Scale (MAS) score ≥ 2
* uncontrolled hypertension, heart problems, infection, or any history of seizure or epilepsy
* neurological disorders that cause motor deficits
* being unable to perform the task or to understand instructions
* presence of pacemaker, pregnancy, cognitive impairment, or psychiatric disorders

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08-09 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Box and block test | baseline (T0), pre-intervention after 1 week of baseline (T1), after 5 weeks of intervention (T2), and at 4 weeks post-intervention (T3)
  Change of box and block test scores

SECONDARY OUTCOMES:
Fugl-Meyer assessment of the upper extremity (FMA) | baseline (T0), pre-intervention after 1 week of baseline (T1), after 5 weeks of intervention (T2), and at 4 weeks post-intervention (T3)
  Change of FMA scores
Jebsen Taylor Hand Function Test (JTT) | baseline (T0), pre-intervention after 1 week of baseline (T1), after 5 weeks of intervention (T2), and at 4 weeks post-intervention (T3)
  Change of JTT scores
Grip strength | baseline (T0), pre-intervention after 1 week of baseline (T1), after 5 weeks of intervention (T2), and at 4 weeks post-intervention (T3)
  Change of Grip strength (JAMAR) scores
Stroke Impact Scale (SIS) | pre-intervention after 1 week of baseline (T1), after 5 weeks of intervention (T2)
  Change of SIS scores

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, South Korea